CLINICAL TRIAL: NCT05279755
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalating Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending and Multiple Ascending Doses of Prosetin in Healthy Volunteers and Participants With Amyotrophic Lateral Sclerosis (ALS) With an Optional Open-Label Extended Treatment Period for ALS Participants Who Complete 14 Days of Blinded Treatment
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Single and Multiple Doses of Prosetin in Healthy Volunteers and Participants With ALS
Acronym: PRO-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ProJenX (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-101; CDMRP-AL240175 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs); 2023-507363-20-00 (EU CTIS Number)
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic lateral sclerosis; MAP4K; prosetin
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts A, B, and C of PRO-101 are double-blind, dose escalating portions of the study. Part D is an open-label extension in which no parties are masked and all participants receive the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part A - single dose of placebo (Placebo Comparator): Healthy volunteers were administered a single dose of prosetin-matched placebo oral solution.
  Interventions: Drug: placebo
- Part A - single ascending doses of prosetin (Experimental): Healthy volunteers were administered a single dose of prosetin oral solution at 0.03, 0.06, 0.12, or 0.24 mg/kg.
  Interventions: Drug: prosetin
- Part B - multiple doses of placebo (Placebo Comparator): Healthy volunteers were administered a once-daily dose of prosetin-matched placebo for 14 days.
  Interventions: Drug: placebo
- Part B - multiple ascending doses of prosetin (Experimental): Healthy volunteers were administered a once-daily dose of prosetin at 0.06 or 0.10 mg/kg for 14 days.
  Interventions: Drug: prosetin
- Part C - multiple doses of placebo in participants with ALS (Placebo Comparator): Participants are administered a once-daily dose of prosetin-matched placebo for 14 days.
  Interventions: Drug: placebo
- Part C - multiple ascending doses of prosetin in participants with ALS (Experimental): Participants will be administered a once-daily dose of prosetin at multiple ascending dose levels for 14 days.
  Interventions: Drug: prosetin
- Part D - open-label administration of prosetin in participants with ALS (Experimental): Participants will be administered a once-daily dose of prosetin for up to 52 weeks.
  Interventions: Drug: prosetin

INTERVENTIONS:
Drug: prosetin — oral solution
  Arms: Part A - single ascending doses of prosetin; Part B - multiple ascending doses of prosetin; Part C - multiple ascending doses of prosetin in participants with ALS; Part D - open-label administration of prosetin in participants with ALS
Drug: placebo — oral solution
  Arms: Part A - single dose of placebo; Part B - multiple doses of placebo; Part C - multiple doses of placebo in participants with ALS

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of prosetin in healthy volunteers and participants with ALS.

DETAILED DESCRIPTION:
PRO-101 is a four-part study. Parts A and B, which respectively evaluated the safety, tolerability, and PK of single and multiple ascending doses of prosetin in 48 healthy volunteers, have been completed.

Parts C and D, which are ongoing, will evaluate the effects of prosetin on safety, tolerability, PK, and biomarkers in 24 participants with ALS. Part C is a double-blind, placebo-controlled, multiple ascending dose component of the study, and Part D is an optional 52-week open-label extension available to ALS participants who complete 14 days of dosing in Part C.

ELIGIBILITY:
PRO-101, Parts A and B, were completed in healthy volunteers.

PRO-101, Parts C and D are ongoing in participants with ALS. Key eligibility criteria are summarized below:

Key Inclusion Criteria - Part C

* Adults ≥18 years of age
* Diagnosis of ALS based on the Gold Coast diagnostic criteria
* Slow Vital Capacity (SVC) >50% predicted
* If being concomitantly treated with riluzole and/or locally approved standard of care treatments, the participant must be on a stable dose for at least 30 days prior to screening and throughout the study
* In the opinion of the Investigator, participant is able to swallow liquid in order to ingest the study medication.

Key Exclusion Criteria - Part C

* Active dementia, neurologic diseases other than ALS, or psychiatric illness that in the opinion of the investigator would affect participation in the current study.
* Significant history or clinical manifestation of comorbid disease in any organ system that currently requires active treatment or is likely to require treatment during the study.
* Any episodes of vertigo in the previous 12 months prior to screening.
* Any medical history of seizures, or any clinically significant EEG finding at Screening or at Day -1.
* A diagnosis of cancer or evidence of continued disease within five years before screening. Protocol-specified exceptions may be considered with approval from the Sponsor's Medical Monitor.
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days prior to the first dose of study medication.
* Prior exposure to any stem cell or gene therapies (investigational or off-label) for the treatment of ALS.

Key Inclusion Criteria- Part D

Participants who meet all of the following criteria may be included in Part D of the study:

* Participants must have completed 14 days of blinded treatment in Part C.
* Participants taking approved ALS standard-of-care medications must remain on stable doses through Day 28 of open-label treatment.
* In the judgment of the Investigator, the participant's participation in the open-label portion of the study is medically appropriate

Key Exclusion Criteria- Part D

* Treatment with any other investigational drug or device throughout the duration of the study is excluded, with the exception of any COVID-19 vaccine or treatment with an emergency use authorization.

NOTE: Other protocol-defined Inclusion/Exclusion Criteria may apply. Please contact trials@projenx.com with any questions about eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-02-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Parts A, B, C, D: Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Part A: Up to 28 days; Part B: Up to 42 days; Part C: Up to 28 days; Part D: Up to 54 weeks
Parts A, B, C, D: Number of Participants with Clinically Significant Laboratory Test Abnormalities | Part A: Up to 28 days; Part B: Up to 42 days; Part C: Up to 28 days; Part D: Up to 54 weeks
Parts A, B, C, D: Number of Participants with Clinically Significant Vital Signs Abnormalities | Part A: Up to 28 days; Part B: Up to 42 days; Part C: Up to 28 days; Part D: Up to 54 weeks
Parts A, B, C, and D: Number of Participants with Clinically Significant Electrocardiogram (ECG) Abnormalities | Part A: Up to 28 days; Part B: Up to 42 days; Part C: Up to 28 days; Part D: Up to 54 weeks
Parts A, B, C, and D: Number of Participants with Clinically Significant Physical Examination Abnormalities | Part A: Up to 28 days; Part B: Up to 42 days; Part C: Up to 28 days; Part D: Up to 54 weeks
Parts A, B, C, and D: Number of Participants with Clinically Significant Neurological Examination Abnormalities | Part A: Up to 28 days; Part B: Up to 42 days; Part C: Up to 28 days; Part D: Up to 54 weeks
Parts A, B, C, and D: Number of Participants with Clinically Significant Ophthalmic Examination Abnormalities | Part A: Up to 28 days; Part B: Up to 42 days; Part C: Up to 28 days; Part D: Up to 54 weeks
Parts C and D: Number of Participants with Clinically Significant Electroencephalogram (EEG) Abnormalities | Part C: Up to 28 days; Part D: Up to 54 weeks

SECONDARY OUTCOMES:
Parts A, B, C, and D: Maximum Observed Concentration (Cmax) of Prosetin in Plasma | Part A: Up to 28 days Part B: Up to 42 days Part C: Up to 28 days Part D: Up to 54 weeks
Parts A, B, C, and D: Time to Reach Maximum Observed Concentration (Tmax) of Prosetin in Plasma | Part A: Up to 28 days Part B: Up to 42 days Part C: Up to 28 days Part D: Up to 54 weeks
Parts A, B, C, and D: Area Under the Concentration-Time Curve (AUC) of Prosetin in Plasma | Part A: Up to 28 days Part B: Up to 42 days Part C: Up to 28 days Part D: Up to 54 weeks
Parts A, B, C, and D: Apparent Terminal Elimination Half-life (t1/2) of Prosetin in Plasma | Part A: Up to 28 days Part B: Up to 42 days Part C: Up to 28 days Part D: Up to 54 weeks
Parts A and D: Measure of Concentration of Prosetin in CSF | Part A: Day 1; Part D: Up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Worldwide Clinical Trials Early Phase Services, San Antonio, Texas
- The Neuro - Montréal Neurological Institute-Hospital, Montreal, Quebec, Canada
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thams S, Lowry ER, Larraufie MH, Spiller KJ, Li H, Williams DJ, Hoang P, Jiang E, Williams LA, Sandoe J, Eggan K, Lieberam I, Kanning KC, Stockwell BR, Henderson CE, Wichterle H. A Stem Cell-Based Screening Platform Identifies Compounds that Desensitize Motor Neurons to Endoplasmic Reticulum Stress. Mol Ther. 2019 Jan 2;27(1):87-101. doi: 10.1016/j.ymthe.2018.10.010. Epub 2018 Oct 19. PMID 30446391
- [Background] Bos PH, Lowry ER, Costa J, Thams S, Garcia-Diaz A, Zask A, Wichterle H, Stockwell BR. Development of MAP4 Kinase Inhibitors as Motor Neuron-Protecting Agents. Cell Chem Biol. 2019 Dec 19;26(12):1703-1715.e37. doi: 10.1016/j.chembiol.2019.10.005. Epub 2019 Oct 31. PMID 31676236